CLINICAL TRIAL: NCT00966888
Title: Selective Use of Postoperative Radiotherapy AftEr MastectOmy - SUPREMO
Brief Title: Radiation Therapy or Standard Therapy in Treating Women With Stage II Breast Cancer Who Have Undergone Mastectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: MRC-BIG2-04; CDR0000642751 (Registry Identifier: PDQ (Physician Data Query)); ISRCTN61145589 (Registry Identifier: ISRCTN (International Standard Randomised Controlled Trial Number Register)); EU-20943
Record Dates: First submitted 2009-08-26; First posted 2009-08-27 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2009-08

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

ARMS (2):
- Arm I (Experimental): Beginning 12 weeks after mastectomy or 6 weeks after adjuvant chemotherapy, patients undergo radiotherapy 5 days a week for 3-5 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: radiation therapy
- Arm II (Active Comparator): Patients receive standard of care and observation only.
  Interventions: Procedure: standard follow-up care

INTERVENTIONS:
Procedure: standard follow-up care — No intervention
  Arms: Arm II
Radiation: radiation therapy — Chest wall radiotherapy
  Arms: Arm I

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays or other types of radiation to kill tumor cells. Giving radiation therapy after surgery may kill any tumor cells that remain after surgery. It is not yet known whether radiation therapy is more effective than observation after mastectomy in treating women with stage II breast cancer.

PURPOSE: This randomized phase III trial is studying radiation therapy to see how well it works compared with standard therapy in treating women with stage II breast cancer who have undergone mastectomy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall survival of women at intermediate risk for locoregional recurrence of breast cancer treated with ipsilateral chest wall adjuvant radiotherapy after mastectomy.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Beginning 12 weeks after mastectomy or 6 weeks after adjuvant chemotherapy, patients undergo radiotherapy 5 days a week for 3-5 weeks in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients receive standard of care and observation only. After completion of study therapy, patients are followed up twice in the first year, and then annually for up to 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed unilateral invasive breast cancer

  * pT1, pN1, M0 disease
  * pT2, pN1, M0 disease
  * pT2, pN0 disease with grade III histology and/or lymphovascular invasion
  * Multifocal breast cancer meeting both of the following criteria:

    * Largest discrete tumor ≥ 2 cm if N0
    * Grade III histology and/or lymphovascular invasion
* No bilateral breast cancer
* Axillary node negative status by axillary clearance, axillary node sampling, or sentinel node biopsy

  * Patients with axillary node positive (1-3 positive nodes, including micrometastases* > 0.2 mm and ≤ 2 mm) must have had an axillary node clearance (minimum of 10 nodes removed) performed

    * No more than 3 pathologically involved lymph nodes
  * No internal mammary nodes visible on sentinel node scintigraphy in the absence of negative histology NOTE: *Isolated tumor cells not counted as micrometastases
* Underwent total mastectomy (with minimum of 1 mm margin clear of invasive cancer and DCIS) and axillary surgery with staging procedure

  * Must have undergone adjuvant systemic chemotherapy if indicated for intermediate-risk breast cancer
  * Patients undergoing immediate breast reconstruction allowed
* No known BRCA1 and BRCA2 carriers
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Not pregnant
* Fit for adjuvant chemotherapy, adjuvant endocrine therapy, and post-operative radiotherapy
* No prior or concurrent malignancy except curatively treated nonmelanomatous skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent trastuzumab
* No prior neoadjuvant systemic therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3500 (Estimated)
Dates: Start 2006-01; Primary Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival
Acute and late morbidity

SECONDARY OUTCOMES:
Chest wall recurrence
Regional recurrence
Disease-free survival
Metastasis-free survival
Cause of death (breast cancer, or intercurrent disease [cardiovascular or non-cardiovascular])
Quality of life
Cost effectiveness

CONTACTS AND LOCATIONS:
Overall Officials: Ian H. Kunkler, MD, Principal Investigator — Edinburgh Cancer Centre at Western General Hospital
Locations (2):
- United Kingdom (2):
  - Edinburgh Cancer Centre at Western General Hospital, Edinburgh, Scotland
  - Royal Infirmary - Castle, Glasgow, Scotland